CLINICAL TRIAL: NCT02158143
Title: A Single High-dose Oral Supplement of Vitamin D in Young Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Hui Wang, Principal Investigator, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-KY1301
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

ARMS (1):
- vitamin D3 (Experimental)
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3

SUMMARY:
evaluated the effect and safety of a single high dose of cholecalciferol in Chinese young people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, younger, Chinese Hans aged from 25-35 years, including 25 and 35 years;
* haven't taken vitamin D supplement for the past 6 months;
* with a normal BMI (18-25 kg/m2);
* with baseline serum 25(OH)D < 30 ng/ml;
* be willing to follow the instruction and complete the study.

Exclusion Criteria:

* clinically diagnosed cardiovascular disease, gastrointestinal disease, endocrine, blood, liver, lung, kidney, nerve or mental illness;
* self-reported current use of any dietary supplements containing vitamin D within the 6 months before enrollment;
* Severe anemia (hemoglobin concentration < 70 g/L);
* Serum 25(OH)D ≥ 30 ng/mL at enrollment;
* participating in other research studies within the 3 months before enrollment;
* history of drug dependence or drug abuse;
* History of heavy drinking (drinking 14 cups or more per week, equivalent to 360 mL beer or 150 mL white wine or 45 mL liquor per cup) and smokers (more than 10 cigarette per day);
* clinical abnormal of blood biochemistry, hematology or urine laboratory values;
* current pregnancy or lactation.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D3 supplementation on serum 25(OH)D changes | within 140 day after supplementation
Effect of vitamin D3 supplementation on serum PTH | within 140 day after supplementation
Effect of vitamin D3 supplementation on serum calcium | within 140 day after supplementation
Effect of vitamin D3 supplementation on serum creatinine | within 140 day of supplementation
Effect of vitamin D3 supplementation on urinary calcium / creatinine | within 140 day after supplementation

SECONDARY OUTCOMES:
Effect of vitamin D3 supplementation on fasting blood glucose | within 140 day after supplementation
Effect of vitamin D3 supplementation on serum lipids | within 140 day after supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Nutrition Sciences, Chinese Academy of Sciences, Shanghai, Shanghai Municipality, China